CLINICAL TRIAL: NCT01656369
Title: Comparative Study Between Delorme Operation With or Without Postanal Repair and Levatorplasty in Treatment of Complete Rectal Prolapse.
Brief Title: Comparative Study Between Delorme Operation With or Without Postanal Repair in Treatment of Complete Rectal Prolapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ayman El Nakeeb, mansoura university, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Rectal prolapse
Record Dates: First submitted 2012-07-26; First posted 2012-08-03 (Estimated); Last update posted 2015-11-23 (Estimated); Status verified 2007-01

CONDITIONS: Rectal Prolapse
Keywords: Delorme operation,incontinence
MeSH Terms: conditions — Rectal Prolapse

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group I delorme operation only. (Active Comparator): A circumferential incision was made in the rectal mucosa approximately 1 cm away from the dentate line. Using electrocautery, the mucosa was stripped to the apex of the prolapse. The muscular layers of the rectal wall were reduced as the mucosa was stripped. Mucosal stripping continued past the apex of the prolapse and then continued inside the prolapsed segment to a point internally that is equivalent to the point of the initial mucosal incision. The underling muscle was plicated by vicryl 2/0.The muscle bite was taken longitudinally from 8 sides to reach a horizontal line of plication at the end. The mucosa was then reanastomosed. Postoperatively, minimal pain medication was required. Early ambulation was encouraged, and patients' diets were advanced as tolerated.
  Interventions: Procedure: Group I: delorme operation only.
- delorme operation with post anal repair (Active Comparator): In group II : post anal repair was added by making transverse incision 7cm behind the anal canal.dissection of intersphincteric plain,plication of internal sphincter by using 3/0 vicryl.The levator ani and external sphincter were then sutured to each other by vicryl 2/0 behind the anal canal followed by skin closure without drain.
  Interventions: Procedure: delorme operation with post anal repair

INTERVENTIONS:
Procedure: Group I: delorme operation only. — A circumferential incision was made in the rectal mucosa approximately 1 cm away from the dentate line. Using electrocautery, the mucosa was stripped to the apex of the prolapse. The muscular layers of the rectal wall were reduced as the mucosa was stripped. Mucosal stripping continued past the apex of the prolapse and then continued inside the prolapsed segment to a point internally that is equivalent to the point of the initial mucosal incision. The underling muscle was plicated by vicryl 2/0.The muscle bite was taken longitudinally from 8 sides to reach a horizontal line of plication at the end. The mucosa was then reanastomosed.
  Other Names: Group I
  Arms: Group I delorme operation only.
Procedure: delorme operation with post anal repair — In group II : post anal repair was added by making transverse incision 7cm behind the anal canal.dissection of intersphincteric plain,plication of internal sphincter by using 3/0 vicryl.The levator ani and external sphincter were then sutured to each other by vicryl 2/0 behind the anal canal followed by skin closure without drain.
  Other Names: Group II
  Arms: delorme operation with post anal repair

SUMMARY:
The aim of the study is to compare Delorme operation alone or with post anal repair and levatorplasty for treating complete rectal prolapse.consecutive patients who were treated for complete rectal prolapse at the Colorectal Surgery Unit were eligible for the study.The patients were randomized into two groups: Group I: consisted of patients were subjected to delorme operation only. Group II: consisted of patients were subjected to delorme operation with post anal repair and levatorplasty.

DETAILED DESCRIPTION:
Rectal procidentia frequently occurs in older women. Patients usually present with obstructed defecation or fecal incontinence. This study is to compare Delorme operation alone or with post anal repair and levatorplasty for treating complete rectal prolapse. Consecutive patients who were treated for complete rectal prolapse at our Colorectal Surgery Unit were eligible for the study. Exclusion criteria include pregnant female, any patients with previous anal surgery, pudendal nerve neuropathy, anal fistula and sepsis or coagulopathy. All patients underwent clinical evaluation, proctoscopic examination, and sigmoidoscopy. Anorectal physiology studies consisted of anal manometry and measurement of pudendal nerve terminal motor latency (PNTML) to exclude pudendal nerve entrapment syndrome. Patients enrolled in the study were randomized into three groups using the closed envelope method. The envelopes were drawn and opened by a nurse not otherwise engaged in the study in the operating room. The patients were randomized into two groups: Group I: consisted of patients were subjected to delorme operation only. Group II: consisted of patients were subjected to delorme operation with post anal repair and levatorplasty.

ELIGIBILITY:
Inclusion Criteria:

* complete rectal prolapse

Exclusion Criteria:

* pregnant female
* any patients with previous anal surgery
* pudendal nerve neuropathy
* anal fistula and sepsis or coagulopathy

Ages: 16 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 82 (Actual)
Dates: Start 2007-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
recurrence rate | one year postoperative
  recurrence rate

SECONDARY OUTCOMES:
changes of bowel habit | early postoperative, after 1 year
  changes of bowel habit
incontinence | 30 day postoperative,and one year postoperative
  incontinence
manometric study | one year postoperative
  manometric study (resting pressure, squeezing pressure)
complications | 30 day postoperative
  stricture, disruption

CONTACTS AND LOCATIONS:
Overall Officials: ayman el nakeeb, MD, Principal Investigator — Mansoura University
Locations (1):
- Ayman El Nakeeb, Al Mansurah, Egypt

REFERENCES:
- [Derived] Youssef M, Thabet W, El Nakeeb A, Magdy A, Alla EA, El Nabeey MA, Fouda el Y, Omar W, Farid M. Comparative study between Delorme operation with or without postanal repair and levateroplasty in treatment of complete rectal prolapse. Int J Surg. 2013;11(1):52-8. doi: 10.1016/j.ijsu.2012.11.011. Epub 2012 Nov 24. PMID 23187047
- See also: Mansoura university — http://www.mans.edu.eg/